CLINICAL TRIAL: NCT00482482
Title: The Safety and Effectiveness of Yoga as Augmentation in Improving Residual Depressive Symptoms in Unipolar and Bipolar Disorders.
Brief Title: Yoga in Unipolar and Bipolar Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Arun Ravindran, Chief, Division of Mood and Anxiety Disorders, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 308/2006
Record Dates: First submitted 2007-06-01; First posted 2007-06-05 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Bipolar Disorder; Major Depression; Dysthymia
Keywords: Yoga; Bipolar disorder; Major depression; Dysthymia; Randomized
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder, Major; Dysthymic Disorder | interventions — Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga (Experimental): Yoga was offered twice a week for 8 weeks, 1.5 hours per session
  Interventions: Behavioral: Yoga
- Psychoeducation (Active Comparator): Psychoeducation was offered twice a week for 8 weeks, 1.5 hours per session
  Interventions: Behavioral: psychoeducation

INTERVENTIONS:
Behavioral: psychoeducation — on weekly basis for 8 weeks
  Arms: Psychoeducation
Behavioral: Yoga — on weekly basis for 8 weeks
  Arms: Yoga

SUMMARY:
Major depression, chronic depression and bipolar depression are complex and difficult disorders to treat. They are often associated with residual symptoms with significant functional impairment. Yoga has been shown to be beneficial in treating depressive symptoms but without the added risks associated with medication use and has the advantage of high consumer appeal (with likelihood of good compliance). However, it has only been tested in unipolar depression, thus far. Yoga if shown to be effective (as an adjunctive to pharmacotherapy) in improving residual symptoms and decreasing risk of relapse, would be of significant long-term benefit to patients not only with major and chronic depression, but also for those with bipolar disorder.

The aim of the study is to determine the safety and effectiveness of Yoga as an augmentation treatment to pharmacotherapy and in comparison to psychoeducation, in improving residual symptoms of depression over 16 weeks and in prevention of relapse/recurrence of mood episodes over 1 year, in subjects with unipolar and bipolar disorders.

DETAILED DESCRIPTION:
Major depression (particularly recurrent and chronic depression) and bipolar depression remain complex and vexing problems for the clinician. They can be difficult to treat with pharmacotherapy alone and the persistence of residual symptoms (with consequent impact on function) and sub-syndromal symptoms increase the risk of relapse. Psychotherapy and alternative therapies have been explored as adjunctive treatments to pharmacotherapy and have shown efficacy in symptom relief. Complementary therapies, like herbal remedies and yoga, have also shown efficacy, but primarily in unipolar depression.

Yoga is a widely accepted practice that is very accessible and adaptable to different age ranges and levels of physical ability. Yoga, has been shown to be effective in the treatment of major depression and dysthymia in randomized, controlled trials. To date,Yoga has not been investigated in subjects with bipolar disorder.

We would like to replicate current investigative results on yoga and depression in a Canadian sample with unipolar and chronic depression, and would like to extend the literature by investigating its efficacy in bipolar disorder. Could adjunctive Yoga treat sub-syndromal depressive symptoms and thus reduce the risk of relapse in patients with unipolar and bipolar depression? With high consumer desirability, there is general agreement on the need for well-designed, randomized controlled trials examining the efficacy and safety of these interventions in clinical populations.

This is a prospective, assessor-blind, crossover, randomized controlled study, and will be carried out in three phases: 1) 16-week treatment phase, 2) 1 year follow-up phase. Forty patients meeting DSM-IV-TR diagnostic criteria for either Major Depression, Dysthymia, Bipolar I or Bipolar II will be recruited. Patients who have provided written consent, have met study criteria, and are stabilized on pharmacotherapy (i.e. receiving either one or two mood stabilizer(s) alone, or in combination with an oral atypical antipsychotic or an antidepressant or lamotrigine) will be enrolled into the study.

All patients will receive treatment with Yoga and psychoeducation in addition to their standard pharmacotherapy and will be randomized to one of two treatment groups groups 1) 8 weeks of yoga followed by 8 weeks of psychoeducation; or 2) 8 weeks of psychoeducation followed by 8 weeks of Yoga. After completion of the treatment phase, there will be a 12-month follow-up phase.

The specific hypotheses are:

1. At week 8 (the end of the first part of the treatment phase), those who are treated with Yoga plus pharmacotherapy would show a decrease in residual depressive symptoms indicated by greater reduction in MADRS scores relative to baseline and an increase in quality of life measures, as compared to those treated with psychoeducation plus pharmacotherapy.
2. At week 16 (the end of the second part of the treatment phase), those who are treated with yoga plus pharmacotherapy would show a decrease in residual depressive symptoms indicated by greater reduction in MADRS scores relative to baseline and an increase in quality of life measures, as compared to those treated with psychoeducation plus pharmacotherapy..
3. Improvement in depressive symptoms will correlate with neuroendocrine changes in salivary cortisol.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients meeting DSM-IV-TR diagnostic criteria for either Major Depression, Dysthymia, Bipolar I or Bipolar II disorder
* MADRS score of ≥10 and ≤24 and a YMRS score of ≤8
* Age 18 to 75 years
* Free of significant physical illness as evidenced by medical history, physical exam, routine clinical investigations and as clinically judged to be able to tolerate physical activities
* Participants taking prophylactic pharmacotherapy for unipolar or bipolar disorders at a stable dose for a minimum of two weeks prior to enrollment

Exclusion Criteria:

* Participants currently in a Manic, Hypomanic, or Mixed Phase
* Participants meeting DSM-IV-TR diagnostic criteria for Rapid Cycling specifier
* History of psychosis not due to Major Depression or Bipolar Disorder, e.g. schizophrenia, schizoaffective disorder, etc.
* Alcohol or Substance Abuse or Dependence within past 3 months
* Participants currently receiving any systematic structured psychotherapy. Supportive therapy is allowed.
* Those with major medical illness, or physical impairment that impact ones ability to participate in the study as evidenced by medical history, physical exam, and clinical investigations

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2007-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | Start of study, 8 weeks and 16 weeks

SECONDARY OUTCOMES:
Salivary cortisol levels | Start of study, 8 weeks, 16 weeks
Clinical Global Impression Scale | Start of study, 8 weeks and 16 weeks
Quality of Life Enjoyment and Satisfaction Scale | Start of study, 8 weeks and 16 weeks
Perceived Stress Scale | Start of study, 8 weeks and 16 weeks
Coping Strategies Scale | Start of study, 8 weeks and 16 weeks
Beck Depression Inventory | Start of study, 8 weeks and 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Arun Ravindran, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addition and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health — http://www.camh.net/research